CLINICAL TRIAL: NCT04101799
Title: Children of Incarcerated Parents - Evaluation of Parental Support Programme in Prison to Promote Positive Parenting and Prevent Children's Ill-health and Delinquency Later in Life
Brief Title: Evaluation of the Parental Support Intervention For Our Children's Sake in Prisons in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Solstickan Foundation, The Sven Jerring Foundation (Unknown)
Responsible Party: Principal Investigator, Åsa Norman, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-04227
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Parenting; Parent-Child Relations
Keywords: Prison; Criminality; Child
MeSH Terms: conditions — Criminal Behavior

STUDY DESIGN:
Intervention Model Description: Controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participating in the For our children's sake intervention, 10 group sessions, 2 hours each
  Interventions: Behavioral: For Our Children's Sake
- Control (Active Comparator): Participating in everyday activities that may include parenting activities in the control prisons
  Interventions: Other: Active control

INTERVENTIONS:
Behavioral: For Our Children's Sake — Parental support with the aim to support positive parenting and promote healthy child development. Conducted in group-format with weekly 2.hour sessions conducted by trained group leaders according to a programme manual.
  Arms: Intervention
Other: Active control — Participating in everyday activities that may include parenting activities in the control prisons
  Arms: Control

SUMMARY:
Evaluation of the effects of the parental support intervention "For our children's sake" on positive parenting outcomes when conducted with incarcerated parents in prisons in Sweden.

DETAILED DESCRIPTION:
Children of incarcerated parents comprise a greatly disadvantaged group in society with elevated risk of ill-health, behavioural problems, and own delinquency and unemployment later in life. Positive parenting comprise an important factor for children's positive and healthy development. Incarcerated parents may have difficulties to engage in positive parenting due to disadvantaged situations affecting parenting negatively such as drug addiction, poverty, or lack of experience of positive parenting in their own childhood. Previous research has suggested that interventions to prevent the intergenerational effect of criminality should be targeting family factors where positive parenting has been emphasised. Internationally developed parenting interventions for incarcerated parents suggest an impact on parenting outcomes such as positive parent-child interaction, parenting knowledge, empathy, parent stress, increased child contact and active parenting, However, the majority of the programmes evaluated to date have been conducted in the US, with a prison and probation context with limited generalisability to the Swedish system. In Sweden, the parenting programme for incarcerated parents, "For our children's' sake" (FOCS) was developed in 2012-2014 with the aim to support positive parenting for the child's healthy development and is currently delivered in Swedish prisons. The aim of this project is to evaluate the effects of the FOCS parenting programme on parenting outcomes through a controlled trial with a parallel implementation process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Serving a sentence at any of the included prisons
* Having at least one child in the ages between 0-18 years. Parents of children aged 0-2 and 13-18 years will not be included in the primary outcome measure, as the measure is not developed for these age groups. These parents will be included in the mediator measurements.
* Are in contact with their child/children in any form. If not, these parents are included in the mediator measurements, as the primary outcome: relationship quality, is not applicable.
* Having the legal right to contact the child
* Not committed either a crime against the child or any violent crime against the other parent

Exclusion Criteria:

* Not fulfilling inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
7-items sub-scale Closeness in the Child Parent Relationship Scale | Positive change in mean score of all 7 items between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at mid-intervention to investigate mediated effects, and a 3-month post intervention follow-up.
  Parent-reported quality in relationship between parent and child on a 5-point scale ('complete agree' to 'completely disagree')

SECONDARY OUTCOMES:
Contact frequency and type between parent and child | Change in mean score of items between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at a 3-month post intervention follow-up.
  Parent-reported frequency (weekly, monthly, less, no contact) and type (letter, telephone, visit/permission, other
Eight items chosen from the sub-scale antisocial intent in the Measures of Criminal Attitudes and Associates scale | Change in mean score of items between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at a 3-month post intervention follow-up.
  Parental attitude to criminality self-reported on a 5-point scale ('complete agree' to 'completely disagree')
Parent interest in other treatment programmes in prison | Change in item score between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at a 3-month post intervention follow-up.
  One item self-reported on an 11-point scale (0 no interest, 10 very high interest)

OTHER OUTCOMES:
14 item parenting attitude from the The Adult-Adolescent Parenting Inventory (AAPI-2) | Change in mean score of items between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at mid-intervention to investigate mediated effects, and a 3-month post intervention follow-up.
  Intermediate outcome/mediator self-reported on a 5-point scale ('complete agree' to 'completely disagree')
6 items parental self-efficacy scale | Change in mean score of items between baseline (pre-intervention) and end of intervention, after 10 weeks. Measurements will also be conducted at mid-intervention to investigate mediated effects, and a 3-month post intervention follow-up.
  Intermediate outcome/mediator self-reported on a 5-point scale ('complete agree' to 'completely disagree')

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Norman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data cannot be shared publicly because of ethical reasons, where public availability would compromise participant privacy. Data are available from the Department of Clinical Neuroscience, Karolinska Institute (contact via registrator@cns.ki.se) for researchers who meet the criteria for access to confidential data.
Supporting Information: Study Protocol
Time Frame: After article publication
Access Criteria: Data cannot be shared publicly because of ethical reasons, where public availability would compromise participant privacy. Data are available from the Department of Clinical Neuroscience, Karolinska Institute (contact via registrator@cns.ki.se) for researchers who meet the criteria for access to confidential data.

REFERENCES:
- [Derived] Norman A, Enebrink P. Effects of a parental support intervention for parents in prison on child-parent relationship and criminal attitude-The For Our Children's Sake pragmatic controlled study. PLoS One. 2023 Mar 23;18(3):e0283177. doi: 10.1371/journal.pone.0283177. eCollection 2023. PMID 36952468
- [Derived] Norman A, Enebrink P. Evaluation of the For Our Children's Sake intervention, parental support in prison to influence positive parenting: study protocol for a controlled trial. BMJ Open. 2020 Jun 7;10(6):e034834. doi: 10.1136/bmjopen-2019-034834. PMID 32513881